CLINICAL TRIAL: NCT05294146
Title: Pharmacokinetic Study With a Loading Dose of Clofazimine in Adult Patients With Nontuberculous Mycobacterial Disease
Acronym: C-LOAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: C-LOAD
Record Dates: First submitted 2022-03-01; First posted 2022-03-24 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2022-09

CONDITIONS: Nontuberculous Mycobacterial Diseases
Keywords: Pulmonary and extrapulmonary NTM diseases
MeSH Terms: interventions — Clofazimine

STUDY DESIGN:
Intervention Model Description: All participants will receive a loading dose regimen of 300 mg clofazimine (CFZ) once daily for 4 weeks and will then continue with a standard dose of 100 mg CFZ once daily until a total 4 months of treatment with CFZ.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Loading dose Clofazimine (Experimental): All participants will receive an (experimental) oral loading dose regimen of 300 mg clofazimine (CFZ) once daily (= 3 capsules of 100 mg) for 4 weeks. Afterwards, all participants will continue with a standard oral dose of 100 mg clofazimine once daily (= 1 capsule of 100 mg) until a total 4 months of treatment with CFZ.
  Interventions: Drug: Clofazimine

INTERVENTIONS:
Drug: Clofazimine — All participants will receive an (experimental) oral loading dose regimen of 300 mg clofazimine once daily (= 3 capsules of 100 mg) for 4 weeks. Afterwards, all participants will continue with a standard oral dose of 100 mg clofazimine once daily (= 1 capsule of 100 mg) until a total 4 months of treatment with CFZ.
  Blood samples will be taken at Day 28 (+/- 2 days), Day 29 (Day 28 +1) and after 4 months of treatment to assess the pharmacokinetics of CFZ, both with the loading dose and the standard dose. In addition, the safety/tolerability of CFZ will monitored.
  Other Names: Lamprene

SUMMARY:
Clofazimine (CFZ) is a promising drug for the treatment of NTM diseases. CFZ is highly active in vitro against M. abscessus and M. avium, the most common NTM pathogens, and shows synergy with macrolides and amikacin. The results from limited clinical studies with CFZ-based treatment regimens are promising. CFZ is currently considered an alternative drug for patients with M. avium complex infections, who are intolerant of first-line drugs. CFZ is a first-line oral drug for treatment of M. abscessus infections.

CFZ might prove to be a cornerstone in NTM treatment, but its optimal dosage is not known. The current dose for adults is 100 mg oncedaily. However, due to the complex pharmacokinetics (PK) of CFZ - it is highly protein bound, extremely lipophilic and accumulates in fatty tissues resulting in a long elimination half-life of ~30 days - it takes several months before steady state, and presumably effective, concentrations are achieved. With the use of a loading dose regimen concentrations similar to those at steady state could be reached faster, possibly leading to improved early treatment efficacy.

The overarching aim of this study is to contribute to dose optimization of CFZ in the treatment of NTM diseases. It will be an explorative, single-center, one-arm, open label, pharmacokinetic study. A number of 10 patients with pulmonary or extrapulmonary NTM disease will be included. Patients will receive a loading dose regimen of 300 mg once daily for 4 weeks and will then continue with a standard dose of 100 mg once daily until a total 4 months of treatment with CFZ.

The primary objective of this study is to describe the PK of CFZ, after 4 weeks of treatment with a loading dose regimen of 300 mg once daily, in adult patients with pulmonary or extrapulmonary NTM disease

ELIGIBILITY:
Inclusion Criteria:

* The participant is diagnosed with pulmonary or extrapulmonary NTM disease and is eligible for treatment with CFZ
* The participant is at least 18 years of age
* The participant has a body weight (in light clothing and with no shoes) of at least 45 kg
* The participant is able and willing to provide written, informed consent

Exclusion Criteria:

* The participant is in poor general condition where participation in the study cannot be accepted per discretion of the Investigator
* There is evidence showing the participant has clinically significant metabolic, gastrointestinal, or other abnormalities that could possibly alter the PK of CFZ
* The participant is diagnosed with cystic fibrosis
* The participant has a prolongation of the QTc interval, > 450 milliseconds for males and > 460 milliseconds for females, on the screening ECG
* The participant has abnormal alanine aminotransferase (ALT) and/or aspartate transferase (AST) levels of > 3 times the upper limit of the laboratory reference range at screening
* The participant is pregnant or is using inadequate contraceptive measures (if applicable)
* The participant is breastfeeding (if applicable)
* The participant has a known or suspected, current drug or alcohol abuse, that is, in the opinion of the Investigator, sufficient to compromise the safety or cooperation of the patient
* The participant has as history of allergy/hypersensitivity to CFZ
* The participant has received clofazimine in the past 3 months before inclusion with the exception of short-term use of no more than 7 days in the period of 1 to 3 months before inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-02-14 (Actual); Primary Completion 2023-05-01 (Actual); Study Completion 2023-08-08 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of clofazimine after a loading dose regimen (1) | 24 hours sampling at Day 28 (+/- 2 days)
  The area under the curve (AUC0-24), after a loading dose regimen of 300 mg once daily for 4 weeks in adult patients with pulmonary or extrapulmonary NTM disease.
Pharmacokinetic parameters of clofazimine after a loading dose regimen (2) | 24 hours sampling at Day 28 (+/- 2 days)
  The peak plasma concentration (Cmax), after a loading dose regimen of 300 mg once daily for 4 weeks in adult patients with pulmonary or extrapulmonary NTM disease.
Pharmacokinetic parameters of clofazimine after a loading dose regimen (3) | 24 hours sampling at Day 28 (+/- 2 days)
  The plasma trough concentration (Cmin), after a loading dose regimen of 300 mg once daily for 4 weeks in adult patients with pulmonary or extrapulmonary NTM disease.

SECONDARY OUTCOMES:
Difference between the highest measured concentrations of CFZ in this study and a reference study | After approximately 1 and 4 months of treatment
  Difference between the highest measured concentrations of CFZ in this study and a reference study (PERC study; EudraCT number 2015-003786-28) after approximately 1 and 4 months of treatment.
The predicted time (e.g. weeks) needed to reach steady state concentrations with and without a loading dose | Expected: 1 to 4 months
  Based on the PK parameters in this study and a reference study (PERC study; EudraCT number 2015-003786-28), the time (in weeks or months) that is needed to reach steady concentrations will be predicted. This will be done for both the loading dose regimen and for a standard dose regimen (i.e. the current clinical care). The goal is to assess how much faster steady state concentrations are reached with a loading dose regimen compared to the standard dose.
Predicted PK parameters (1) | After approximately 1 and 4 months of treatment
  The predicted area under the curve (AUC0-24), after approximately 1 and 4 months of treatment in both this study and a reference study (PERC study; EudraCT number 2015-003786-28)
Predicted PK parameters (2) | After approximately 1 and 4 months of treatment
  The predicted peak concentration (Cmax), after approximately 1 and 4 months of treatment in both this study and a reference study (PERC study; EudraCT number 2015-003786-28)
Predicted PK parameters (3) | After approximately 1 and 4 months of treatment
  The predicted trough concentration (C0), after approximately 1 and 4 months of treatment in both this study and a reference study (PERC study; EudraCT number 2015-003786-28)
Adverse Events | Through study completion, a period of 4 months
  The number of (participants with) adverse events will be measured. Adverse events will be graded according to the 'Common Terminology Criteria for Adverse Events' (CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. R.E. Aarnoutse, PharmD, PhD, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboud university medical center, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Stemkens R, Lemson A, Koele SE, Svensson EM, Te Brake LHM, van Crevel R, Boeree MJ, Hoefsloot W, van Ingen J, Aarnoutse RE. A loading dose of clofazimine to rapidly achieve steady-state-like concentrations in patients with nontuberculous mycobacterial disease. J Antimicrob Chemother. 2024 Dec 2;79(12):3100-3108. doi: 10.1093/jac/dkae309. PMID 39378281